CLINICAL TRIAL: NCT07120958
Title: What Impact Does Uterine Immunity Have on the Success of Euploid Thawed Embryos?
Brief Title: The Impact of Uterine Immunity and Its Alterations on the Embryo Implantation Process
Acronym: UTIMEE
Status: Enrolling by invitation | Type: Observational
Sponsor: Momo Fertilife (Other)
Collaborators: University of Bari (Other); University of Florence (Other); Casa Sollievo della Sofferenza-IRCCS, San Giovanni Rotondo (Unknown)
Responsible Party: Principal Investigator, Daniele Ferri, IVF Lab Manager, Momo Fertilife
Other Study IDs: 32/cf/2025
Record Dates: First submitted 2025-07-25; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Infertility Assisted Reproductive Technology
Keywords: interleukin; ngs; art; icsi; implantation; euploid; uterine immunity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Endometrial biopsy stored at -80 C°
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- endometrial biopsy with pregnancy
- endometrial biopsy without pregancy

SUMMARY:
Evaluation of uterine immunity, histological picture, and endometrial microbiome for embryo implantation

ELIGIBILITY:
Inclusion Criteria:

Female patients aged >18 and <43 years at the time of embryo transfer.

Transfer of cryopreserved embryos diagnosed as euploid through preimplantation genetic testing for aneuploidy (PGT-A).

Embryo transfer performed at the blastocyst stage.

Exclusion Criteria:

Patients with an intrauterine device (IUD) in situ within the three months prior to study enrollment.

Presence of autoimmune diseases and/or ongoing treatment with corticosteroids.

Structural or pathological abnormalities of the uterine cavity, including but not limited to polyps, intramural myomas measuring 2-4 cm, submucosal fibroids, uterine septum, or hydrosalpinx, identified during study participation. Patients with a history of these conditions may be included if the pathology has been resolved prior to the initiation of any study-related procedures or sample collection.

Presence of severe or uncontrolled fungal or viral infections which, in the opinion of the principal investigator, may compromise the patient's ability to participate or affect the integrity of study outcomes.

Any medical condition or illness that is unstable, poses a potential risk to patient safety, or may interfere with adherence to the study protocol.

Patients lacking a confirmed preimplantation genetic diagnosis of euploidy.

Patients with a clinical diagnosis of endometriosis or adenomyosis.

Ages: 20 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women who undertake ART treatment in South Italy
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Characterise the molecular immunologic mechanism underlying embryo implantation | from enrollment to the pregnancy test (12 days after embryo transfer)
  The main objective of this research is to characterise the molecular immunologic mechanism underlying embryo implantation. These outcomes will be assessed regarding the percentage of expressivity of some interleukins in pregnant couples and those who are not

SECONDARY OUTCOMES:
to study the possible correlations of the expression of the interleukins involved in the implantation process of the embryo | The endometrial biopsy on which the interleukin dosage will be done, will be taken one month before the embryo transfer
  to study the possible correlations of the expression of the interleukins involved with related anatomical and histological pictures. Interleukin dosage will be assessed through PCR. The unit of measure is ng/ml.

OTHER OUTCOMES:
to assess whether progesterone levels can alter the immune response | the same day of the embryo transfer
  immunofluorescence device; unit of measure: ng/ml

CONTACTS AND LOCATIONS:
Overall Officials: Domenico Baldini, Degree in Medicine and Surgery, Principal Investigator — Momo Fertilife
Locations (1):
- MOMO' Fertilife, Bisceglie, BT, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nagaeva O, Jonsson L, Mincheva-Nilsson L. Dominant IL-10 and TGF-beta mRNA expression in gammadeltaT cells of human early pregnancy decidua suggests immunoregulatory potential. Am J Reprod Immunol. 2002 Jul;48(1):9-17. doi: 10.1034/j.1600-0897.2002.01131.x. PMID 12322898
- [Background] Vitoratos N, Papadias C, Economou E, Makrakis E, Panoulis C, Creatsas G. Elevated circulating IL-1beta and TNF-alpha, and unaltered IL-6 in first-trimester pregnancies complicated by threatened abortion with an adverse outcome. Mediators Inflamm. 2006;2006(4):30485. doi: 10.1155/MI/2006/30485. PMID 17047289
- [Background] Lombardelli L, Logiodice F, Kullolli O, Haller H, Agostinis C, Bulla R, Rukavina D, Piccinni MP. At Embryo Implantation Site IL-35 Secreted by Trophoblast, Polarizing T Cells towards IL-35+ IL-10+ IL-4+ Th2-Type Cells, Could Favour Fetal Allograft Tolerance and Pregnancy Success. Int J Mol Sci. 2022 Apr 28;23(9):4926. doi: 10.3390/ijms23094926. PMID 35563316
- [Background] Ledee N, Petitbarat M, Prat-Ellenberg L, Dray G, Cassuto GN, Chevrier L, Kazhalawi A, Vezmar K, Chaouat G. The uterine immune profile: A method for individualizing the management of women who have failed to implant an embryo after IVF/ICSI. J Reprod Immunol. 2020 Nov;142:103207. doi: 10.1016/j.jri.2020.103207. Epub 2020 Sep 14. PMID 32971456
- [Background] Szekeres-Bartho J. The Role of Progesterone in Feto-Maternal Immunological Cross Talk. Med Princ Pract. 2018;27(4):301-307. doi: 10.1159/000491576. Epub 2018 Jun 27. PMID 29949797
- [Background] Piccinni MP, Raghupathy R, Saito S, Szekeres-Bartho J. Cytokines, Hormones and Cellular Regulatory Mechanisms Favoring Successful Reproduction. Front Immunol. 2021 Jul 28;12:717808. doi: 10.3389/fimmu.2021.717808. eCollection 2021. PMID 34394125
- [Background] Mahajan D, Kumar T, Rath PK, Sahoo AK, Mishra BP, Kumar S, Nayak NR, Jena MK. Dendritic Cells and the Establishment of Fetomaternal Tolerance for Successful Human Pregnancy. Arch Immunol Ther Exp (Warsz). 2024 May 23;72(1). doi: 10.2478/aite-2024-0010. eCollection 2024 Jan 1. PMID 38782369
- [Background] Zhou J, Yan P, Ma W, Li J. Cytokine modulation and immunoregulation of uterine NK cells in pregnancy disorders. Cytokine Growth Factor Rev. 2025 Feb;81:40-53. doi: 10.1016/j.cytogfr.2024.11.007. Epub 2024 Nov 23. PMID 39603954
- [Background] Parasar P, Guru N, Nayak NR. Contribution of macrophages to fetomaternal immunological tolerance. Hum Immunol. 2021 May;82(5):325-331. doi: 10.1016/j.humimm.2021.02.013. Epub 2021 Mar 11. PMID 33715911
- [Background] Wang W, Sung N, Gilman-Sachs A, Kwak-Kim J. T Helper (Th) Cell Profiles in Pregnancy and Recurrent Pregnancy Losses: Th1/Th2/Th9/Th17/Th22/Tfh Cells. Front Immunol. 2020 Aug 18;11:2025. doi: 10.3389/fimmu.2020.02025. eCollection 2020. PMID 32973809
- [Background] Szekeres-Bartho J. Immunological relationship between the mother and the fetus. Int Rev Immunol. 2002 Nov-Dec;21(6):471-95. doi: 10.1080/08830180215017. PMID 12650238
- [Background] Abu-Raya B, Michalski C, Sadarangani M, Lavoie PM. Maternal Immunological Adaptation During Normal Pregnancy. Front Immunol. 2020 Oct 7;11:575197. doi: 10.3389/fimmu.2020.575197. eCollection 2020. PMID 33133091